CLINICAL TRIAL: NCT00358592
Title: Randomized Controlled Trial of the Efficacy of the Mobius ™ Retractor in Performing Cesarean Sections in Patients With BMI ≥35kg/m2
Brief Title: Comparison of Tissue Retractors During Cesarean Delivery in Obese Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: Apple Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06C.78
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Cesarean Section; Obesity
Keywords: surgical instruments; cesarean section; obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Device: Mobius™ retractor
Device: traditional metal retraction instruments

SUMMARY:
This is a randomized controlled trial comparing the use of the Mobius™ retractor to the use of traditional metal retraction instruments in non-urgent cesarean deliveries of obese women. The Mobius™ retractor was designed for abdominal surgery to improve visualization of the surgical field through standard surgical incisions and is now a standard instrument used for cesarean deliveries at Thomas Jefferson University Hospital. We hypothesize that the use of the Mobius™ retractor during cesarean deliveries in obese women decreases operative time, blood loss, number of transfusions, infectious morbidity, incision length, and intra- / post-operative antiemetic and pain medication use, while increasing surgeon satisfaction.

DETAILED DESCRIPTION:
The Mobius™ retractor has been used in many obese cesarean deliveries based on the theory that it provides superior visualization. There have been no clinical trials to determine if this "added" exposure offers any measurable significant benefits to justify the added cost. This study will determine if the Mobius™ retractor does provide a measurable difference in outcomes, compared to the traditional retraction instruments.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women undergoing non-urgent cesarean delivery

Exclusion Criteria:

* women undergoing urgent cesarean delivery
* BMI <35kg/m2
* women undergoing vaginal delivery
* positive urine drug screen or known history of methadone maintenance or substance abuse

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-07; Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
operative time

SECONDARY OUTCOMES:
blood loss
number of transfusions
infectious morbidity
incision length
intra and postoperative antiemetic medication use
intra and postoperative pain medication use
surgeon satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Jason K Baxter, MD, MSCP, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States